CLINICAL TRIAL: NCT01381445
Title: A Randomised, Double-blind (for GW870086), Placebo-controlled Study of Topical GW870086 Formulation to Explore the Potential for Skin Thinning in Healthy Adult Volunteers
Brief Title: A Study Assessing GW870086's Potential to Cause Skin Thinning
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 113435
Record Dates: First submitted 2011-06-16; First posted 2011-06-27 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Clobetasol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GW870086 0.2% & GW870086 2% (Experimental): GW870086 0.2%, 2% & placebo each applied to an identified area for 42 days.
  Interventions: Drug: GW870086 0.2%; Drug: GW870086 2%; Drug: Placebo
- GW870086 2% & Clobetasol Propionate (Experimental): GW870086 2% & placebo applied to an identified area for 42 days, while Clobetasol Propionate is applied to an area for 21 days
  Interventions: Drug: GW870086 2%; Drug: Clobetasol Propionate; Drug: Placebo

INTERVENTIONS:
Drug: GW870086 0.2% — White to slightly coloured opaque cream
  Arms: GW870086 0.2% & GW870086 2%
Drug: GW870086 2% — White to slightly coloured opaque cream
Drug: Clobetasol Propionate — White cream
  Arms: GW870086 2% & Clobetasol Propionate
Drug: Placebo — White to slightly coloured opaque cream

SUMMARY:
This study is a randomised, double-blind, placebo-controlled study of topical GW870086 to explore the potential for skin thinning in healthy adult volunteers after 42±2 days of treatment. Twenty (20) healthy volunteers will be randomised to receive placebo and GW870086 2% cream, they will also receive either of the following treatments: GW870086 0.2% cream, or clobetasol propionate 0.05% cream.

DETAILED DESCRIPTION:
This study is a randomised, double-blind, placebo-controlled study of topical GW870086 to explore the potential for skin thinning in healthy adult volunteers after 42±2 days of treatment. The primary objective of this study is to assess the thickness of the skin using ultrasound. The secondary objectives are to assess skin thinning using a visual scale for skin atrophy and telangiectasia, safety and tolerability of GW870086 and to assess the pharmacokinetics of GW870086 administered as a cream for 42±2 days.

Twenty (20) healthy volunteers will be randomised to receive placebo and GW870086 2% cream. They will also receive either of the following treatments: GW870086 0.2% cream, or clobetasol propionate 0.05% cream. Subjects will apply all 3 treatments once daily during the 42±2 day treatment period. However subjects who are randomised to receive the unblinded clobetasol propionate will only apply this once daily for a maximum of 21±2 days but will continue to dose with the other 2 treatments. If significant evidence of skin thinning is observed in any of the treatment arms (25% reduction in skin thickness measured using ultrasound) then application of this treatment will be discontinued. Three areas of approximately 5 x 5 cm on the arm will be identified and each treatment will be applied to the same area throughout the 42±2 day treatment period.

ELIGIBILITY:
Inclusion Criteria:

* AST (Aspartate aminotransferase), ALT (Alanine aminotransferase), alkaline phosphatase and bilirubin ≤ 1.5xULN (Upper limit of normal)(isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Healthy as determined by an experienced physician.
* Male or female between 18 and 55 years of age inclusive.
* A female subject is eligible to participate if she is of:

  • Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the protocol contraception methods if they wish to continue their HRT during the study.
* Male subjects with female partners of child-bearing potential must agree to use one of the protocol contraception methods.
* BMI within the range 19.0 - 29.0 kg/m2 (inclusive).
* Capable of giving written informed consent.
* Single QTc, QTcB < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.

Exclusion Criteria:

* Any sign of weak or fragile skin, striae, or similar, in the areas which will be evaluated.
* Tattoos or body art on the upper arms.
* Foreseeable intensive UV exposure during the study (solar or artificial). Subjects must not be exposed to direct sunlight or skin tanning devices (e.g. sunbed) for the duration of the study.
* A positive pre-study test for Hepatitis B or Hepatitis C antibody within 3 months of screening.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities.
* A positive pre-study drug/alcohol screen.
* A positive test for HIV (Human Immunodeficiency Virus) antibody.
* History of regular alcohol consumption within 6 months of the study.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications or components thereof.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* Subjects who are kept due to regulatory or juridical order in an institution.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Consumption of red wine, Seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-04-14 (Actual); Primary Completion 2011-07-07 (Actual); Study Completion 2011-07-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in skin thickness using ultrasound between GW870086 (0.2% and 2%) versus placebo | Days; 1, 14, 21, 28, 42, 43

SECONDARY OUTCOMES:
Clinical evaluation of treated skin areas using assessment of clinical signs and symptoms according to the visual scores of skin atrophy and telangiectasia | Days; 7, 14, 21, 28, 35, 42, 43
The assessment of safety parameters; adverse events, clinical laboratory tests, ECG, and vital signs | 6 weeks
Plasma concentrations of GW870086 | Days 14 & 42
Cmax of GW870086 | Days 14 & 42
Tmax of GW870086 | Days 14 & 42
AUC of GW870086 | Days 14 & 42

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 113435 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/113435?search=study&study_ids=113435#rs
- Available data/document: Informed Consent Form: 113435 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113435 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113435 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113435 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113435 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113435 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113435 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register